CLINICAL TRIAL: NCT03393182
Title: A Multicenter Randomized Controlled Trial Comparing the Quality of Life Between Laparoscopy-assisted Distal Gastrectomy and Totally Laparoscopic Distal Gastrectomy for Gastric cancer_KLASS 07 (CKLASS01)(Korea-China Collaborated Study)
Brief Title: Comparing the Quality of Life Between LADG and TLDG for Gastric Cancer_KLASS07 (CKLASS01)).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Shanghai Medical College of Fudan University (Unknown)
Responsible Party: Principal Investigator, Sungsoo Park, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KLASS07(CKLASS01)
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Quality of Life; Gastric Cancer; Surgery; Surgical Complication
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, multi-center trial that comparing surgical complications and Quality of Life between "Totally laparoscopic distal gastrectomy" and "Laparoscopy-assisted distal gastrectomy" in Korea.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TLDG arm (Experimental): TLDG arm(Totally laparoscopic distal gastrectomy)
  : After lymphadenectomy, gastrectomy and reconstruction procedure are performed intracorporeally without mini-laparotomy.
  Interventions: Procedure: TLDG arm
- LADG arm (Experimental): LADG arm(Laparoscopy-assisted distal gastrectomy)
  : After lymphadenectomy, gastrectomy and reconstruction procedure are performed through mini-laparotomy
  Interventions: Procedure: LADG arm

INTERVENTIONS:
Procedure: TLDG arm — After lymphadenectomy, gastrectomy and reconstruction procedure are performed intracorporeally without mini-laparotomy(TLDG)
  Arms: TLDG arm
Procedure: LADG arm — After lymphadenectomy, gastrectomy and reconstruction procedure are performed extracorporeally through mini-laparotomy(LADG)
  Arms: LADG arm

SUMMARY:
The present randomized study is designed to compare the quality of life between the patients undergoing laparoscopy-assisted and totally laparoscopic distal gastrectomy for gastric cancer, and therefore to evaluate the superiority of totally laparoscopic distal gastrectomy to laparoscopy-assisted distal gastrectomy.

DETAILED DESCRIPTION:
The primary endpoint of this trial is the early postoperative morbidity, that is defined as complications that occur within 30 days after surgery.

Early postoperative morbidity is classified as follows:

(1) wound morbidity (2) surgical site morbidity: anastomosis bleeding or leakage, duodenal stump leakage, postoperative bleeding, afferent loop or efferent loop obstruction, etc.; (3) lung morbidity: atelectasis, pleural effusion, empyema, pneumothorax, etc.; (4) intestinal obstruction morbidity (5) urinary tract morbidity (6) intra-abadominal abscess (7) postoperative pancreatitis (8) pancreatic fistula (9) intestinal fistula 10) others: lymphorrhea, diarrhea, etc.

The secondary end point is the questionnaire score regarding QOL. This is assessed by the Korean versions of the EORTC QLQ-C30 (version 3.0) and STO22 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proven gastric adenocarcinoma (by preoperative gastrofiberscopy)
* Age between 20 and 80 years old
* Eastern Cooperative Oncology Group performance statu of 0 or 1
* Clinical stage IA (T1N0M0) or IB (T1N1M0 / T2N0M0) according to the 7th edition of the American Joint Committee on Cancer system10 (Clinical stage was determined based on the finding of gastrofiberscopy and abdominal computed tomography)
* Scheduled for laparoscopic distal gastrectomy with D1+ or D2 lymphadenectomy, and possible for R0 surgery by this procedures (Lymphadenectomy is performed on the basis of the criteria of the Japanese Gastric Cancer Treatment Guidelines 2010 (ver.3).)
* Patients who gave a consent and signed the formal paper permitted by Institutional Review Board (IRB) after hearing a full description of the study (purpose and contents) prior to the participation

Exclusion Criteria:

* Patients who received stomach surgery (i.e. gastrectomy or gastrojejunostomy) in the past
* Patients with intraabdominal adhesion due to previous intraperitoneal surgery
* Patients who recently diagnosed with gastric cancer and received either anticancer treatment or radiation therapy
* Patients who requires combined organ resection due to aggression of gastric cancer or other diseases
* Patients who received surgeries due to primary cancer of other organs, or had anticancer treatment or radiation therapy in the last five years (patients whose skin basal cell carcinoma and insitu cervical cancer are completely cured are exceptions).
* Vulnerable people who can't communicate or are pregnant (or planning to be pregnant)
* Patients who are currently participating or participated in other clinical trials in the last six months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Postoperative 30-day morbidity rate | Postoperative 30-day
  Check the morbidity rate
  :Wound, seroma, hematoma, wound infection, wound dehiscence, wound evisceration, Fluid collection/Abscess, Intraabdominal bleeding, Intraluminal bleeding, Postoperative ileus, Anastomosis stenosis, Anastomosis leakage, Pancreatitis or pancreatic fistula, Complication(Pulmonary, Urinary, Renal, Hepatic, Cardiac, Endocrine) etc.

SECONDARY OUTCOMES:
QOL measurement : EORTC QLQ-C30/STO22 | screening(pre op) / Postoperative 30-day,3-month,6-month,12-month
  EORTC QLQ-C30/STO22

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang Y, Li Z, Tian Y, Yu J, Wang J, Lee C, Wang K, He X, Qiao Q, Ji G, Xu Z, Yang L, Xu H, Du X, Su X, Xing J, Niu Z, Zhu L, Yan S, Li Y, Wang J, Li Z, Zhao Y, You J, Jing C, Fan L, Du Y, Zhao G, Song W, Xuan Y, Zang M, Chen J, Park S, Huang H; China-Korea Laparoscopic Gastrointestinal Surgery Study (CKLASS) Cooperative Group. Morbidity and quality of life of totally laparoscopic versus laparoscopy-assisted distal gastrectomy for early gastric cancer: a multi-center prospective randomized controlled trial (CKLASS01). Gastric Cancer. 2025 Jan;28(1):131-144. doi: 10.1007/s10120-024-01561-y. Epub 2024 Nov 5. PMID 39499377
- [Derived] Lee HH, Lee CM, Lee MS, Jeong IH, Son MW, Kim CH, Yoo MW, Oh SJ, Son YG, Choi SI, Jung MR, Seo SH, Park SH, Hwang SH, Min JS, Park S. Morbidity and Mortality After Laparoscopy-Assisted Distal Gastrectomy and Totally Laparoscopic Distal Gastrectomy to Treat Gastric Cancer: An Interim Report: A Phase III Multicenter, Prospective, Randomized Trial (The KLASS-07 Trial). J Gastric Cancer. 2024 Jul;24(3):257-266. doi: 10.5230/jgc.2024.24.e22. PMID 38960885
- [Derived] Park SH, Lee CM, Hur H, Min JS, Ryu SW, Son YG, Chae HD, Jeong O, Jung MR, Choi CI, Song KY, Lee HH, Kim HG, Jee YS, Hwang SH, Lee MS, Kim KH, Seo SH, Jeong IH, Son MW, Kim CH, Yoo MW, Oh SJ, Kim JG, Hwang SH, Choi SI, Yang KS, Huang H, Park S. Totally laparoscopic versus laparoscopy-assisted distal gastrectomy: the KLASS-07: a randomized controlled trial. Int J Surg. 2024 Aug 1;110(8):4810-4820. doi: 10.1097/JS9.0000000000001543. PMID 38716987
- [Derived] Lee CM, Park JH, In Choi C, Lee HH, Min JS, Jee YS, Jeong O, Chae H, Choi SI, Huang H, Park S. A multi-center prospective randomized controlled trial (phase III) comparing the quality of life between laparoscopy-assisted distal gastrectomy and totally laparoscopic distal gastrectomy for gastric Cancer (study protocol). BMC Cancer. 2019 Mar 7;19(1):206. doi: 10.1186/s12885-019-5396-8. PMID 30845995